CLINICAL TRIAL: NCT01323972
Title: Consistency of Immunogenicity and Non Inferiority of Three Production Lots of GSK Biologicals' Candidate Malaria Vaccine in Children
Brief Title: Consistency of Immunogenicity and Non Inferiority of GSK Biologicals' Candidate Malaria Vaccine Lots in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 113398
Record Dates: First submitted 2011-02-24; First posted 2011-03-28 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2017-10

CONDITIONS: Malaria
Keywords: Malaria; Plasmodium falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- GSK 257049-Lot 1 Group (Experimental): Healthy male or female children aged 5 to 17 months received 3 doses of the GSK 257049 vaccine from the commercial scale lot 1 (formulation 1 of the GSK 257049 vaccine) administered intramuscularly (IM) in the deltoid of the left arm, at Day 0, at Month 1 and at Month 2.
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine (257049)
- GSK 257049-Lot 2 Group (Experimental): Healthy male or female children aged 5 to 17 months received 3 doses of the GSK 257049 vaccine, from the commercial scale lot 2 (formulation 2 of the GSK 257049 vaccine) administered intramuscularly (IM) in the deltoid of the left arm, at Day 0, at Month 1 and at Month 2.
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine (257049)
- GSK 257049-Lot 3 Group (Experimental): Healthy male or female children aged 5 to 17 months received 3 doses of the GSK 257049 vaccine, from the commercial scale lot 3 (formulation 3 of the GSK 257049 vaccine) administered intramuscularly (IM) in the deltoid of the left arm, at Day 0, at Month 1 and at Month 2.
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine (257049)
- GSK 257049-Pilot Group (Experimental): Healthy male or female children aged 5 to 17 received 3 doses of the GSK 257049 vaccine from the pilot scale (pilot formulation of the GSK 257049 vaccine) administered intramuscularly (IM) in the deltoid of the left arm, at Day 0, at Month 1 and at Month 2.
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine (257049)

INTERVENTIONS:
Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine (257049) — 4 different lots of the candidate malaria vaccine (257049) representative of either commercial (manufacturing) process or pilot plant process

SUMMARY:
The purpose of this study is to show the consistency of different lots of a candidate vaccine (257049) against malaria developed by GlaxoSmithKline (GSK) Biologicals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol.
* A male or female child between, and including, 5 and 17 months of age at the time of the first vaccination.
* Signed or thumb-printed informed consent obtained from the parent(s)/LAR(s) of the child. Where parent(s)/LAR(s) are illiterate, the consent form will be countersigned by a witness.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects who have received three documented doses of hepatitis B vaccine.

Exclusion Criteria:

* Same sex twins.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures.
* Moderate or severe malnutrition at screening defined as weight for age Z-score less than 2.
* Acute disease and/or fever at the time of enrolment
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or medical history.
* Use of a drug or vaccine that is not approved for that indication other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/administration of a licensed vaccine not foreseen by the study protocol within 7 days of the first dose of study vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Administration of immunoglobulins and/or any blood products within 1 month preceding the first dose of study vaccine or planned administration during the study period.
* Child in care.
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial.

Ages: 5 Months to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 327 (Actual)
Dates: Start 2011-05-16 (Actual); Primary Completion 2011-11-22 (Actual); Study Completion 2012-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Nigeria (2):
  - GSK Investigational Site, Enugu
  - GSK Investigational Site, Jos

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 113398 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113398 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113398 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113398 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113398 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113398 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 327 subjects originally enrolled, 7 dropped out of the study before receiving the first vaccination.
Period: Overall Study
Arm/Group | GSK 257049-Lot 1 Group | GSK 257049-Lot 2 Group | GSK 257049-Lot 3 Group | GSK 257049-Pilot Group
Started | 81 | 79 | 80 | 80
Completed | 79 | 76 | 78 | 79
Not Completed | 2 | 3 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Migrated/moved from study area | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK 257049-Lot 1 Group | GSK 257049-Lot 2 Group | GSK 257049-Lot 3 Group | GSK 257049-Pilot Group | Total
Number analyzed (Participants) | 81 | 79 | 80 | 80 | 320
Age, Continuous [Mean (Standard Deviation); unit: Months] | 9.8 (3.35) | 10.2 (3.56) | 10.1 (3.24) | 10.2 (3.01) | 10.07 (3.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 40 | 33 | 30 | 147
  Male | 37 | 39 | 47 | 50 | 173
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 81 | 79 | 80 | 80 | 320

OUTCOME MEASURES:

1. Primary Outcome: Anti-Circumsporozoite (Anti-CS) Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs) and are measured in titers.
Time Frame: One month post-dose 3 (Month 3)
Population: The analyses were performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- GSK 257049-Pooled Group: This is a pooled group, made up of GSK 257049-Lot 1 Group, GSK 257049-Lot 2 Group and GSK 257049-Lot 3 Group.
Arm/Group | GSK 257049-Lot 1 Group | GSK 257049-Lot 2 Group | GSK 257049-Lot 3 Group | GSK 257049-Pooled Group | GSK 257049-Pilot Group
Number analyzed (Participants) | 72 | 72 | 73 | 217 | 72
Titers | 319.6 [268.9 to 379.8] | 241.4 [207.6 to 280.7] | 302.3 [259.4 to 352.3] | 285.8 [260.7 to 313.3] | 271.7 [228.5 to 323.1]
Statistical Analysis 1: Comparison: GSK 257049-Lot 1 Group vs GSK 257049-Lot 2 Group; Demonstration of the lot-to-lot consistency between GSK 257049-Lot 1 and GSK 257049-Lot 2 in terms of anti-Circumsporozoite (anti-CS) immunogenicity; Test type: Other; GMT ratio = 1.32, 95% CI 2-sided [1.06 to 1.65] — Consistency was demonstrated if one month post Dose 3, the 2-sided 95% confidence interval (CI) of the geometric mean titer (GMT) ratio between all pairs of lots were within [0.5, 2]
Statistical Analysis 2: Comparison: GSK 257049-Lot 1 Group vs GSK 257049-Lot 3 Group; Demonstration of the lot-to-lot consistency between GSK 257049-Lot 1 and GSK 257049-Lot 3 in terms of anti-Circumsporozoite (anti-CS) immunogenicity; Test type: Other; GMT ratio = 1.06, 95% CI 2-sided [0.85 to 1.32] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GSK 257049-Lot 2 Group vs GSK 257049-Lot 3 Group; Demonstration of the lot-to-lot consistency between GSK 257049-Lot 2 and GSK 257049-Lot 3 in terms of anti-Circumsporozoite (anti-CS) immunogenicity; Test type: Other; GMT ratio = 0.8, 95% CI [0.64 to 1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GSK 257049-Pooled Group vs GSK 257049-Pilot Group; Demonstration of non-inferiority of the commercial scale lots of GSK 257049 to the pilot scale lot in terms of anti-Circumsporozoite (anti-CS) immunogenicity; Test type: Non-Inferiority — Non-inferiority was demonstrated if one month post Dose 3, the upper limit (UL) of the 2-sided 95% CI of the GMT ratio of the pilot scale lot (Control Group) over the pooled commercial scale lots (Pooled Log Group) was below 2; GMT ratio = 0.95, 95% CI [0.79 to 1.15]

2. Secondary Outcome: Anti-hepatitis B (Anti-HB) Antibody Concentrations
Description: Antibody concentrations are presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL).
Time Frame: One month post-dose 3 (Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK 257049-Lot 1 Group | GSK 257049-Lot 2 Group | GSK 257049-Lot 3 Group | GSK 257049-Pooled Group | GSK 257049-Pilot Group
Number analyzed (Participants) | 72 | 72 | 73 | 217 | 72
mIU/mL | 54250.2 [43293.6 to 67979.7] | 46067.3 [33919.2 to 62566.2] | 67384.7 [52271.4 to 86867.7] | 55273.5 [47508.3 to 64308.0] | 74105.0 [58613.6 to 93690.7]

3. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: Over a 7-day (Days 0-6)post-vaccination period after each dose and across doses
Population: The analyses were performed on the Total Vaccinated cohort, which included all vaccinated subjects with their symptom sheets filled in, for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 257049-Lot 1 Group | GSK 257049-Lot 2 Group | GSK 257049-Lot 3 Group | GSK 257049-Pilot Group
Number analyzed (Participants) | 81 | 79 | 80 | 80
Participants
  Any Pain, Dose 1 | 16 | 14 | 15 | 13
  Grade 3 Pain, Dose 1 | 0 | 0 | 0 | 0
  Any Redness, Dose 1 | 4 | 1 | 1 | 4
  Grade 3 Redness, Dose 1 | 0 | 0 | 0 | 0
  Any Swelling, Dose 1 | 4 | 2 | 3 | 3
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Any Pain, Dose 2 | 7 | 4 | 4 | 8
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Grade 3 Pain, Dose 2 | 0 | 0 | 0 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Any Redness, Dose 2 | 1 | 1 | 1 | 3
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 | 0
  Any Swelling, Dose 2 | 1 | 1 | 1 | 3
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Any Pain, Dose 3 | 4 | 2 | 4 | 3
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Grade 3 Pain, Dose 3 | 0 | 0 | 0 | 0
  Any Redness, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Any Redness, Dose 3 | 3 | 2 | 2 | 1
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Grade 3 Redness, Dose 3 | 0 | 0 | 0 | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Any Swelling, Dose 3 | 3 | 3 | 2 | 1
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Grade 3 Swelling, Dose 3 | 0 | 0 | 0 | 0
  Any Pain, Across Doses | 27 | 20 | 20 | 22
  Grade 3 Pain, Across Doses | 0 | 0 | 0 | 0
  Any Redness, Across Doses | 8 | 4 | 4 | 7
  Grade 3 Redness, Across Doses | 0 | 0 | 0 | 0
  Any Swelling, Across Doses | 8 | 6 | 6 | 6
  Grade 3 Swelling, Across Doses | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination. Grade 3 loss of appetite = not eating at all. Grade 3 irritability = crying that could not be comforted/prevented normal activity. Grade 3 drowsiness = drowsiness that prevented normal activity. Grade 3 fever = fever higher than (>) 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Over a 7-day (Days 0-6) post-vaccination period after each dose and across doses
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 257049-Lot 1 Group | GSK 257049-Lot 2 Group | GSK 257049-Lot 3 Group | GSK 257049-Pilot Group
Number analyzed (Participants) | 81 | 79 | 80 | 80
Participants
  Any Drowsiness, Dose 1 | 1 | 0 | 0 | 0
  Related Drowsiness, Dose 1 | 0 | 0 | 0 | 0
  Grade 3 Drowsiness, Dose 1 | 0 | 0 | 0 | 0
  Any Irritability, Dose 1 | 3 | 0 | 3 | 0
  Related Irritability, Dose 1 | 0 | 0 | 0 | 0
  Grade 3 Irritability, Dose 1 | 0 | 0 | 0 | 0
  Any Loss of appetite, Dose 1 | 4 | 4 | 1 | 3
  Related Loss of appetite, Dose 1 | 0 | 0 | 1 | 0
  Grade 3 Loss of appetite, Dose 1 | 0 | 0 | 0 | 0
  Any Fever, Dose 1 | 25 | 23 | 27 | 24
  Related Fever, Dose 1 | 11 | 8 | 11 | 5
  Grade 3 Fever, Dose 1 | 0 | 0 | 1 | 0
  Any Drowsiness, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Any Drowsiness, Dose 2 | 2 | 1 | 1 | 3
  Related Drowsiness, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Related Drowsiness, Dose 2 | 1 | 0 | 0 | 0
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Grade 3 Drowsiness, Dose 2 | 0 | 0 | 0 | 0
  Any Irritability, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Any Irritability, Dose 2 | 4 | 1 | 4 | 7
  Related Irritability, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Related Irritability, Dose 2 | 2 | 0 | 2 | 3
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Grade 3 Irritability, Dose 2 | 0 | 0 | 0 | 0
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Any Loss of appetite, Dose 2 | 5 | 1 | 1 | 5
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Related Loss of appetite, Dose 2 | 1 | 0 | 0 | 0
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Grade 3 Loss of appetite, Dose 2 | 0 | 0 | 0 | 0
  Any Fever, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Any Fever, Dose 2 | 28 | 17 | 24 | 20
  Related Fever, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Related Fever, Dose 2 | 11 | 7 | 9 | 7
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 81 | 78 | 79 | 80
  Grade 3 Fever, Dose 2 | 0 | 0 | 2 | 0
  Any Drowsiness, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Any Drowsiness, Dose 3 | 3 | 2 | 2 | 1
  Related Drowsiness, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Related Drowsiness, Dose 3 | 0 | 0 | 0 | 0
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Grade 3 Drowsiness, Dose 3 | 0 | 0 | 0 | 0
  Any Irritability, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Any Irritability, Dose 3 | 6 | 3 | 4 | 3
  Related Irritability, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Related Irritability, Dose 3 | 3 | 1 | 2 | 2
  Grade 3 Irritability, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Grade 3 Irritability, Dose 3 | 0 | 0 | 0 | 0
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Any Loss of appetite, Dose 3 | 3 | 2 | 2 | 1
  Related Loss of appetite, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Related Loss of appetite, Dose 3 | 0 | 0 | 0 | 0
  Grade 3 Loss of appetite, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Grade 3 Loss of appetite, Dose 3 | 0 | 0 | 0 | 0
  Any Fever, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Any Fever, Dose 3 | 23 | 10 | 21 | 19
  Related Fever, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Related Fever, Dose 3 | 15 | 6 | 15 | 10
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 80 | 78 | 78 | 80
  Grade 3 Fever, Dose 3 | 1 | 0 | 1 | 0
  Any Drowsiness, Across doses | 6 | 3 | 3 | 3
  Related Drowsiness, Across doses | 1 | 0 | 0 | 0
  Grade 3 Drowsiness, Across doses | 0 | 0 | 0 | 0
  Any Irritability, Across doses | 12 | 4 | 10 | 9
  Related Irritability, Across doses | 5 | 1 | 4 | 5
  Grade 3 Irritability, Across doses | 0 | 0 | 0 | 0
  Any Loss of appetite, Across doses | 11 | 7 | 4 | 7
  Related Loss of appetite, Across doses | 1 | 0 | 1 | 0
  Grade 3 Loss of appetite, Across doses | 0 | 0 | 0 | 0
  Any Fever, Across doses | 49 | 41 | 47 | 41
  Related Fever, Across doses | 27 | 19 | 27 | 18
  Grade 3 Fever, Across doses | 1 | 0 | 3 | 0

5. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within the 30-day (Days 0-29) post-vaccination period
Population: The analyses were performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 257049-Lot 1 Group | GSK 257049-Lot 2 Group | GSK 257049-Lot 3 Group | GSK 257049-Pilot Group
Number analyzed (Participants) | 81 | 79 | 80 | 80
Participants | 63 | 60 | 70 | 58

6. Secondary Outcome: Number of Subjects With Serious Adverse Events
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Up to 8 months post-dose 1
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 257049-Lot 1 Group | GSK 257049-Lot 2 Group | GSK 257049-Lot 3 Group | GSK 257049-Pilot Group
Number analyzed (Participants) | 81 | 79 | 80 | 80
Participants | 6 | 5 | 12 | 4

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 7-day (Days 0-6) post-vaccination period. Unsolicited AEs: during the 30-day (Days 0-29) post-vaccination period. SAEs: during the entire study period (Day 0 - Month 8).
Arm/Group | GSK 257049-Lot 1 Group | GSK 257049-Lot 2 Group | GSK 257049-Lot 3 Group | GSK 257049-Pilot Group
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/79 | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 6/81 | 5/79 | 12/80 | 4/80
Other Adverse Events (participants affected / at risk) | 77/81 | 71/79 | 71/80 | 67/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK 257049-Lot 1 Group (N=81) | GSK 257049-Lot 2 Group (N=79) | GSK 257049-Lot 3 Group (N=80) | GSK 257049-Pilot Group (N=80)
Bronchopneumonia (Infections and infestations) | 4 | 2 | 6 | 1
Malaria (Infections and infestations) | 4 | 4 | 4 | 1
Tonsillitis (Infections and infestations) | 0 | 3 | 3 | 0
Sepsis (Infections and infestations) | 2 | 1 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Pneumonitis chemical (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK 257049-Lot 1 Group (N=81) | GSK 257049-Lot 2 Group (N=79) | GSK 257049-Lot 3 Group (N=80) | GSK 257049-Pilot Group (N=80)
Malaria (Infections and infestations) | 36 | 35 | 41 | 33
Respiratory tract infection (Infections and infestations) | 27 | 23 | 27 | 23
Upper respiratory tract infection (Infections and infestations) | 18 | 19 | 23 | 16
Gastroenteritis (Infections and infestations) | 8 | 12 | 7 | 8
Diarrhoea (Gastrointestinal disorders) | 9 | 3 | 2 | 7
Bronchopneumonia (Infections and infestations) | 3 | 3 | 8 | 2
Enteritis (Gastrointestinal disorders) | 7 | 5 | 5 | 3
Furuncle (Infections and infestations) | 4 | 5 | 5 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 5 | 2 | 1
Pain (General disorders) | 27 | 20 | 20 | 22
Redness (General disorders) | 8 | 4 | 4 | 7
Swelling (General disorders) | 8 | 6 | 6 | 6
Drowsiness (General disorders) | 6 | 3 | 3 | 3
Irritability (General disorders) | 12 | 4 | 10 | 9
Loss of appetite (General disorders) | 11 | 7 | 4 | 7
Fever (axillary) (General disorders) | 49 | 41 | 47 | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.